CLINICAL TRIAL: NCT04769726
Title: Evaluation of Pre-meal Load of Raw Almonds on Postprandial Hyperglycemia and Other Metabolic Responses in Asian Indians With Prediabetes
Brief Title: Pre-meal Load of Raw Almonds and Postprandial Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NDOC/11/2017
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Intervention
Keywords: almonds; Asian Indians; Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): premeal load of almonds
  Interventions: Dietary Supplement: almonds
- control (No Intervention): standard diet

INTERVENTIONS:
Dietary Supplement: almonds — almond intervention (20 g) before three major meals (60g per day) for 3 days in subacute phase, before OGTT in the acute phase ad for 3 months in chronic phase
  Arms: treatment

SUMMARY:
A few studies show the effect of almonds on postprandial hyperglycemia (PPHG); high blood glucose after meals. In our previous study on intervention with almonds, we observed a significant decrease in HbA1C and a small decrease in fasting blood glucose indicating a possible effect of almonds on PPHG. Studies have shown that a preload of a food article that is high in protein, mono-unsaturated fatty acids, fiber, and low in carbohydrates, such as almonds could be helpful in stimulating insulin secretion and help improve postprandial hyperglycemia. The proposed study shall be undertaken to assess the effect of almond supplementation on postprandial hyperglycemia in Asian Indians with prediabetes.

DETAILED DESCRIPTION:
* Acute Phase Study: Randomized controlled cross over study design Number of arms: 2, almond and control, n=60 needed (30 in each arm) Subjects randomized to almonds arm are given a preload of 20 g of almonds 30 minutes prior to ingestion of 75 g of glucose, while those in the control arm do not have any food/almonds before OGTT. Blood samples are collected at (minutes): -30, 30, 0, 30, 60, 90 and 120. Cross over of these subjects is done and OGTT repeated in a similar manner. Assessment of blood glucose, serum insulin, glucagon, C-peptide, serum triglycerides, free fatty acids, DPP-IV, and GLP1 levels are done at these time points.
* Sub-Acute Study:

Three-day almond preload study monitored with CGMS, n=60 needed. All study participants undergoing OGTT are further studied with CGMS for three days each and then crossed over. Those in almonds arm continue to receive preload of almonds (20g almonds, 30 minutes before breakfast, lunch and dinner)for three days and then studied without almond preload after cross over. A washout period of 7 days separates cross-over period.

o Chronic Phase Study: Ninety days almond preload study monitored with self-monitoring of blood glucose; n=60 needed.

This is a randomized controlled parallel-arm study to evaluate the long-term effect of preload of almonds on hyperglycemia. Subjects fulfilling the inclusion/exclusion criteria are randomized to either the control arm or the almond arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Prediabetes as diagnosed on oral glucose tolerance test (OGTT): Fasting blood glucose ≥100mg/dl and <126 mg/dl and 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75 gram anhydrous oral glucose) or 2-h plasma glucose

  * 140mg/dl and <200mg/dl alone.

Exclusion Criteria:

* Acute infections and advanced end-organ damage
* History of hepatitis or pancreatitis, abnormal liver and renal functions
* Recent (<3 months) changes in weight (≥5%) and/or weight changing medications
* Any known allergy to nuts
* uncontrolled hypertension or hypothyroidism
* suffering from acute infection or any debilitating disease or with renal failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose levels [AUC 0-2 hrs on oral glucose tolerance test (OGTT)] | 8 days

SECONDARY OUTCOMES:
postprandial blood glucose levels [AUC 0-4 hrs on continuous glucose monitoring system{CGMS}] | 15 days
Postprandial hyperglycaemia (blood glucose levels 2 hrs post OGTT) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Anoop misra, New Delhi, India

REFERENCES:
- [Derived] Gulati S, Misra A, Tiwari R, Sharma M, Pandey RM, Upadhyay AD, Chandra Sati H. Premeal almond load decreases postprandial glycaemia, adiposity and reversed prediabetes to normoglycemia: A randomized controlled trial. Clin Nutr ESPEN. 2023 Apr;54:12-22. doi: 10.1016/j.clnesp.2022.12.028. Epub 2022 Dec 29. PMID 36963852
- [Derived] Gulati S, Misra A, Tiwari R, Sharma M, Pandey RM, Upadhyay AD, Sati HC. Beneficial effects of premeal almond load on glucose profile on oral glucose tolerance and continuous glucose monitoring: randomized crossover trials in Asian Indians with prediabetes. Eur J Clin Nutr. 2023 May;77(5):586-595. doi: 10.1038/s41430-023-01263-1. Epub 2023 Feb 2. PMID 36732571